CLINICAL TRIAL: NCT01206075
Title: A Pilot Study to Assess the Safety and Efficacy of Mozobil ± G-CSF in Mobilizing Hematopoietic Stem Cells (CD34+ Cells) in Adults With Beta-thalassemia Major
Brief Title: Evaluating the Safety and Effectiveness of Mozobil Mobilization in Adults With Beta-Thalassemia Major
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); George Papanicolaou Hospital (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Thalia Papayannopoulou, Professor, Medicine, Hematology, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36078-B; P01HL053750 (NIH); 2P01HL053750 (NIH)
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Beta-Thalassemia
Keywords: Beta Thalassemia Major; Hematopoietic Stem Cell Mobilization; Gene Transfer Techniques
MeSH Terms: conditions — beta-Thalassemia | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mozobil + G-CSF - 001 (Other): Up to four patients (splenectomized and non-splenectomized) previously mobilized with G-CSF (previous study), who failed to yield by 2 leukaphereses sufficient CD34+ cells for a future gene therapy procedure, will receive the combination of G-CSF+Mozobil
  Interventions: Drug: Mozobil
- Mozobil (Other): Sixteen or more patients (non-splenectomized and splenectomized) who were not previously mobilized will receive Mozobil alone.
  Interventions: Drug: Mozobil
- Mozobil + G-CSF - 002 (Other): Patients who, in this study, fail to mobilize sufficient yields of blood stem cells with Mozobil alone will be invited to be re-mobilized with the combination of Mozobil plus G-CSF.
  Interventions: Drug: Mozobil

INTERVENTIONS:
Drug: Mozobil — Previously mobilized splenectomized patients who failed to yield sufficient numbers of cells with Mozobil alone will receive low doses G-CSF subcutaneously (starting at 2.5µg/kg/day and adjusted to the degree of leukocytosis), and Mozobil at 240µg/kg starting on the 4th or 5th day of G-CSF, followed by one to three leukaphereses. Previously non-splenectomized patients who failed to yield sufficient numbers of cells with Mozobil alone will receive G-CSF at 10µg/kg/day subcutaneously for 4-7 days, and Mozobil at 240µg/kg starting on the 4th or 5th day of G-CSF, followed by one to three leukaphereses.
  Other Names: Plerixafor; AMD 3100
  Arms: Mozobil + G-CSF - 002
Drug: Mozobil — Previously mobilized splenectomized patients who failed to yield sufficient numbers of cells with G-CSF in the previous study will receive low doses G-CSF subcutaneously (starting at 2.5µg/kg/day and adjusted to the degree of leukocytosis), and Mozobil at 240µg/kg starting on the 4th or 5th day of G-CSF, followed by one to three leukaphereses. Previously non-splenectomized patients who failed to yield sufficient numbers of cells with G-CSF in the previous study will receive G-CSF at 10µg/kg/day subcutaneously for 4-7 days, and Mozobil at 240µg/kg starting on the 4th or 5th day of G-CSF, followed by one to three leukaphereses.
  Other Names: Plerixafor; AMD3100
  Arms: Mozobil + G-CSF - 001
Drug: Mozobil — Up to sixteen patients (splenectomized and non-splenectomized) who were not previously mobilized will receive Mozobil at 240µg/kg for one to three days, followed by one to three leukaphereses.
  Other Names: Plerixafor; AMD3100
  Arms: Mozobil

SUMMARY:
Thalassemia is considered the most common genetic disorder worldwide, occurring with high frequency in Mediterranean areas, the Middle East, Southeast Asia, and the Pacific Islands. Currently, the only cure for thalassemia is bone marrow transplantation from a related, compatible donor. Gene transfer, achieved by transplantation of the patient's own blood stem cells that have been genetically-modified with the corrected gene, could potentially cure thalassemia.

The first step in developing gene transfer for treatment of thalassemia is to develop a safe and effective method to obtain blood stem cells from thalassemia patients. Eventually, high numbers of genetically modified cells will need to be infused into the patient for clinical gene transfer to be effective. The blood stem cells are obtained by giving a "mobilization" agent to the patients. This causes the stem cells to leave the bone marrow and go into the blood. The purpose of this study is to test the safety and effectiveness of the new mobilization agent, Mozobil, in causing mobilization of blood stem cells for patients with beta-thalassemia major.

DETAILED DESCRIPTION:
The purpose of this study is to optimize blood stem cell mobilization in adults with beta thalassemia major. We seek a method of mobilization that will be safe, with minimum side effects, and that will yield high numbers of blood stem cells. For successful gene therapy of thalassemia, high numbers of genetically modified stem cells will need to be introduced into the patient. Participants will include beta-thalassemia patients who failed to mobilize sufficiently with G-CSF (in our previous protocol) and new patients. In this study we will focus on the safety and effectiveness of mobilization with Mozobil or with Mozobil plus G-CSF. Following mobilization, blood stem cells will be recovered using leukapheresis, a procedure similar to a blood donation, in which mobilized white blood cells are collected from the blood of the patient.

During drug administration and leukapheresis, patients will be hospitalized at George Papanicolaou Hospital in Thessaloniki, Greece. Patients who failed to mobilize in the previous protocol will receive Mozobil and G-CSF and will be hospitalized for 5-8 days for the duration of drug administration and leukapheresis. They will receive G-CSF for several days; Mozobil will be added on the last few days of G-CSF. New patients will receive Mozobil only and will be hospitalized for 2-3 days for drug administration and leukapheresis. Mozobil is administered at 240µg/kg, under the skin. Participants will undergo two or three leukapheresis procedures in a row if low numbers of blood stem cells were recovered in the first (and possibly second) leukapheresis. Participants will be discharged from the hospital the day following the last leukapheresis procedure. Weekly follow-up visits will occur for the next month, either at G. Papanicolaou Hospital, or at the participant's local doctor's office. The total period of study participation is approximately 5 weeks. In the event that Mozobil alone does not cause mobilization of high levels of blood cells, patients will be invited to repeat the protocol three months later, receiving Mozobil and G-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Βeta- thalassemia major
* Age >18<50
* Karnofsky performance status ³80%
* Splenectomized patients or patients with spleen volume <800cm3 (only for the non splenectomized patients who will receive Mozobil + G-CSF)
* Compliant with regular transfusions and regular chelation
* Liver iron by MRI <280μmol/gr or ³1.7msec by T2*MRI
* Heart iron by MRI >2.8 (SI/SD) or ³9msec by T2*MRI
* Hepatitis B or C virus load negative by PCR (polymerase chain reaction)
* Left ventricular ejection fraction (LVEF) >45% by echocardiogram
* Adequate respiratory function with DLCO >50%
* Negative pregnancy test, if female
* Ability to give informed consent and willingness to meet all the expected requirements of the protocol for the duration of the study

Exclusion Criteria:

* History of thrombosis or known thrombophilia
* Symptomatic viral, bacterial or fungal infection within 6 weeks prior eligibility evaluation
* Pregnancy or lactation
* HIV positivity
* History of malignancy, other than local skin cancer
* Other systematic disease non thalassemia-associated
* Splenectomized patients with platelet count >900,000 (only for the splenectomized patients who will receive low dose G-CSF+ Mozobil)
* Additional risk factors for thrombosis, including Factor V Leiden; antiphospholipid antibodies and less than 50% of the lowest normal value for the following procoagulants: antithrombin 3, protein C, or protein S.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety and effectiveness of Mozobil for mobilization of patients with beta thalassemia major | Five weeks
  i) To determine the safety of peripheral blood stem cell (PBSC) mobilization with Mozobil alone or with Mozobil + G-CSF in adults with b-thalassemia major ii) To collect with Mozobil or Mozobil+G-CSF a total of at least 6 X 10e6 CD34+ cells/kg for a subsequent clinical beta-globin gene transfer trial.

SECONDARY OUTCOMES:
Clonogenic capacity, transducibility, and engraftment potential (in a mouse model) of genetically modified cells | Six months
  Secondary: i)To determine the clonogenic capacity of cells mobilized by Mozobil alone, or by Mozobil + G-CSF, ii) To determine the cells' ability to be transduced with a recombinant lentivirus vector for beta-globin, iii) To determine the transduced cells' potential to engraft in a xenograft model.

CONTACTS AND LOCATIONS:
Overall Officials: Thalia Papayannopoulou, MD, Principal Investigator — University of Washington
Locations (1):
- George Papanicolaou Hospital, Thessaloniki, Greece